CLINICAL TRIAL: NCT01378351
Title: Vestibular Dysfunction as a Cause of Chronic Nausea & Vomiting: A Follow up Study
Brief Title: Vestibular Dysfunction as a Cause of Chronic Nausea & Vomiting: A Follow up Survey
Status: Terminated | Type: Observational
Why Stopped: Inadequate recruitment, investigator left institution
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 011-085
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Dysfunction of Vestibular System; Nausea Persistent; Vomiting
MeSH Terms: conditions — Vomiting | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaire survey — Mailed questionnaire investigating response to empiric treatment trials, further investigations by otolarygology and possible alternative diagnoses.

SUMMARY:
The purpose of this study is to characterize the accompanying symptoms, evaluation and management of patients with chronic vestibular dysfunction presenting with nausea and vomiting.

DETAILED DESCRIPTION:
Based on prior study, a significant portion of patients referred for refractory gastroparesis in fact have signs suggestive of vestibular dysfunction as the cause of chronic nausea and vomiting. Our prior retrospective study identified a population of said subjects.

The aim of this study is to further characterize the concomitant symptoms, course of diagnosis, treatment and long-term follow up (up to 5 yrs) of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of nausea and vomiting for at least 4 weeks
* Abnormal modified Fukuda stepping test on examination (>90 degree rotation from midline while marching in place for 60 seconds) or nystagmus or abnormal Rhomberg test

Exclusion Criteria:

* Pregnancy
* Unable to complete questionnaire survey

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient gastroenterology clinic
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Improvement of nausea and vomiting | 1 to 2 months

SECONDARY OUTCOMES:
Associated symptoms | 1 to 2 months
Alternate diagnoses | 1 to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Schiller, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States